CLINICAL TRIAL: NCT03942159
Title: Modification of the Human Colon and Oral Microbiome by Allogeneic HSCT in Recipients and Correlation With the Microbiome of the Donor
Brief Title: Modification of the Human Colon and Oral Microbiome by Allogenic HSCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Other Study IDs: NCHPOI-2019-01
Record Dates: First submitted 2019-04-29; First posted 2019-05-08 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Human Microbiome; HSCT
Keywords: Microbiome; stem cell transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — colon and oral swab
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Donors: HLA-matched or haploidentical nursing relative donors
- Patients: recipients of allogeneic HSCT

SUMMARY:
Allogenic HSCT brings significant changes in biodiversity and composition of the gut microbiome through antibiotic usage, the mucosal damage due to the chemo- and radiotherapy toxicity; compromised oral nutritional intake and graft-versus-host disease with gut damage as the complication. Aim of the study is to investigate the composition of the microbiota in both recipient and nursing relative donor, reveal changes in biodiversity after HSCT via 3-time points V3V4 16S rRNA and NGS sequencing of the colon and oral swabs, 3-indoxyl-sulfate measurement in the urine.

ELIGIBILITY:
Inclusion Criteria:

* indications to alloHSCT
* nursing healthy donors 3-55 y.o.

Exclusion Criteria:

* unable to give samples for the test
* graft rejection
* previous HSCT

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric recipients and their donors receiving treatment in the Dmitry Rogachev National Medical Research Center Of Pediatric Hematology, Oncology, and Immunology
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2019-05-14 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
beta-index dynamics | 7 days before HSCT
  biodiversity (beta-index) dynamics between time points before and after HSCT
beta-index dynamics | 7 days after HSCT
  biodiversity (beta-index) dynamics between time points before and after HSCT
beta-index dynamics | 60 days after HSCT
  biodiversity (beta-index) dynamics between time points before and after HSCT

SECONDARY OUTCOMES:
Proportion of patients with microbial domination after HSCT | 7 days after HSCT
  evaluation of the dynamics of the microbial domination between time points before and after HSCT
Proportion of patients with microbial domination after HSCT | 60 days after HSCT
  evaluation of the dynamics of the microbial domination between time points before and after HSCT
Shannon-index dynamics | 7 days before HSCT
  biodiversity (Shannon-index - an information statistic index, which means it assumes all species are represented in a sample and that they are randomly sampled) dynamics between time points before and after HSCT
Shannon-index dynamics | 7 days after HSCT
  biodiversity (Shannon-index - an information statistic index, which means it assumes all species are represented in a sample and that they are randomly sampled) dynamics between time points before and after HSCT
Shannon-index dynamics | 60 days after HSCT
  biodiversity (Shannon-index - an information statistic index, which means it assumes all species are represented in a sample and that they are randomly sampled) dynamics between time points before and after HSCT
ROC (receiver operating characteristic)-curve of NGS (new-generation sequence) | 7 days before HSCT
  sensitivity of NGS as a method of biodiversity evaluation
ROC (receiver operating characteristic)-curve of NGS (new-generation sequence) | 7 days after HSCT
  sensitivity of NGS as a method of biodiversity evaluation
ROC (receiver operating characteristic)-curve of NGS (new-generation sequence) | 60 days after HSCT
  sensitivity of NGS as a method of biodiversity evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Michael Maschan, PhD, Principal Investigator — National Research Center for Pediatric Hematology , Moscow, Russian Federation
Locations (1):
- Dmitry Rogachev National Research Center of Pediatric Hematology, Oncology and Immunology, Moscow, Russia